CLINICAL TRIAL: NCT05222737
Title: Quantitave Assessment of Aggregatibacter Actinomycetemcomitans and Porphyromonas Gingivalis by Real -Time PCR Following Application of Diode Laser in Severe Periodontitis (A RANDIOMIZED CONTROLLED CLINICAL TRIAL)
Brief Title: Quantitation of Bacteria Associated With Severe Periodontitis by Real -Time PCR Following Application of Diode Laser
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, amira hafez, Resident at department of periodontolgy. Alexandria university, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lasers in periodontology
Record Dates: First submitted 2022-01-25; First posted 2022-02-03 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Active Comparator): intra pocket diode laser application
  Interventions: Device: medency diode laser
- control group (Active Comparator): antibiotic adminstration
  Interventions: Drug: spirazole forte

INTERVENTIONS:
Device: medency diode laser — intra pocket application of diode laser
  Arms: test group
Drug: spirazole forte — adminstration of spirazole forte with a dose 17 mg per kg
  Arms: control group

SUMMARY:
1. Primary objective To measure the gingival crevicular levels of A.actinomycetemcomitans and P.gingivalis after intra-pocket application of diode laser in severe periodontitis (stage 3 grade C) patients.
2. Secondary objective To compare the levels of the same microorganisms as in cases of diode laser therapy to those after conventional treatment with systemic antibiotic administration in severe periodontitis (stage 3 grade C) patients.
3. to measure clinical parameters probing depth,attachment loss and mobility grade

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes having severe periodontitis (stage 3 grade C) with interdental clinical attachment loss (CAL) ≥ 5.
2. Patients' age between 15 and 35 years old with rapid bone loss showed by radiograph.
3. Systemically healthy patients.
4. Radiographic bone loss extending to middle or apical third of root.
5. Probing depth (PD) ≥ 6 mm.

Exclusion Criteria:

1. Use of antibiotics during the last 3 months.
2. Pregnancy.
3. Any systemic condition that might affect the study.
4. Use of mouthwash containing antimicrobials during the previous 3 weeks.
5. Smoking.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Quantitation of Aggrecatibacter .actinomycetemcomitans and porphyromonas gingivalis bacteria | baseline
  To measure the gingival crevicular levels of A.actinomycetemcomitans and P.gingivalis after intra-pocket application of diode laser in severe periodontitis(stage 3 grade C) patients

SECONDARY OUTCOMES:
comparing levels of bacteria between test and control groups | baseline
  To compare the levels of the same microorganisms as in cases of diode laser therapy to those after conventional treatment with systemic antibiotic administration in severe periodontitis ( stage 3 grade C) patients.

OTHER OUTCOMES:
Probing depth(PPD) | Baseline ,one month and 3 months
  Measure PPD at baseline and after treatment
Clinical Attachment loss(CAL) | Baseline ,one month and 3 months
  Measure CAL at baseline and after treatment
Mobility grade | Baseline ,one month and 3 months
  Measure mobility grade at baseline and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hafez, Alexandria, Egypt

REFERENCES:
- [Derived] Anwar SK, Hafez AM, Roshdy YS. Clinical and microbiological efficacy of intra-pocket application of diode laser in grade C periodontitis: a randomized controlled clinical trial. BMC Oral Health. 2024 Feb 23;24(1):270. doi: 10.1186/s12903-024-04031-0. PMID 38395824